CLINICAL TRIAL: NCT02234037
Title: A Pilot Study of Physical Conditioning and Decitabine for Newly Diagnosed AML Patients Age ≥ 60 Who Are Not Candidates for Standard Induction Chemotherapy
Brief Title: Physical Conditioning and Decitabine for Newly Diagnosed AML Patients Age ≥ 60
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Martha Arellano, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00064866; WINSHIP2381-12 (Other: Winship Cancer Institute)
Record Dates: First submitted 2014-02-27; First posted 2014-09-09 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia | interventions — Decitabine; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine and Exercise (Experimental): 8-week program of physical conditioning and decitabine treatment in newly diagnosed AML patients ≥ 60 years of age who are not candidates for standard induction chemotherapy.
  Interventions: Drug: Decitabine; Behavioral: Exercise

INTERVENTIONS:
Drug: Decitabine — Decitabine will be administered intravenously at dose of 20mg/m² on 5 consecutive days every 28 days (1 cycle = 28 days) for a total of 2 cycles according to standard practice. Cycle 2 will proceed on time despite cytopenias, given that patients are not expected to be in remission after only 1 cycle of decitabine.
  Other Names: Dacogen
Behavioral: Exercise — Each patient will participate in 2-3 exercise sessions per week supervised by a physical therapist. Each exercise session will comprise > 10 minutes of muscle strengthening, > 10 minutes of aerobic exercise (treadmill walking or cycling), > 10 minutes of stretching/range of motion exercises, and up to 10 minutes of individualized functional exercise (determined based on patient's reported deficits/targets in activities of daily living).

SUMMARY:
STUDY BACKGROUND AND PURPOSE:

Acute myelogenous leukemia (AML) is a common type of blood cancer in adults, and is more common with increasing age. AML is harder to treat in older patients, with typically poor responses to standard chemotherapy.

Patients with AML are typically given intensive induction chemotherapy, but many older patients cannot tolerate the side effects of this therapy. Decitabine has been shown to be active and better tolerated in frail patients with AML; however, most patients still relapse.

Recent studies suggest that improving the performance status and fitness of older AML patients prior to induction chemotherapy may help to lessen side effects.

This study will test the combination of decitabine treatment with physical exercise in elderly patients with AML who are not candidates for standard induction chemotherapy.

STUDY DESCRIPTION:

This is a pilot study to test the combination of decitabine treatment with an 8-week physical exercise program in AML patients ≥ 60 years of age who are not candidates for standard induction chemotherapy. Patients who are eligible to take part must give their written agreement before they can be enrolled.

This study will enroll 20 patients who are not candidates for standard induction chemotherapy. Patients will begin an 8-week program of physical exercise, including 2-3 sessions per week supervised by a physical therapist. During this 8-week period, patients will be given 2 cycles of decitabine therapy (daily infusion for 5 consecutive days of a 28-day cycle).

Patients will be followed to assess the safety and tolerability of the program. Patients will also give blood samples that will be used to assess their response to treatment. Patients will be evaluated for their physical fitness before and after the 8-week exercise program and will complete questionnaires to assess their quality of life before and after the program.

DETAILED DESCRIPTION:
Primary Objectives:

• Number of patients age 60 and older with newly diagnosed AML and who are not candidates for standard induction chemotherapy who complete an 8-week program of physical conditioning and decitabine treatment. The goal is set at 30% of 20 enrolled patients completing the 8 weeks of decitabine and physical conditioning program.

Secondary Objectives:

* Number of patients with adverse events as a measure of safety and tolerability of the physical conditioning program during decitabine therapy.
* Number of patients with overall response (complete response, disease-free survival [DFS], and overall survival [OS]) of the rehabilitated patients after conclusion of the 8-week program.
* Changes in quality of life among study subjects before and after the 8-week exercise program.
* Changes in cytokine profiles drawn at baseline, 4 weeks and 8 weeks.

Treatment Plan:

* Twenty subjects, age 60 and older with newly diagnosed AML who are deemed by their referring physicians not to be candidates for standard induction chemotherapy will be recruited from the inpatient and outpatient services at Emory University Hospital and the Winship Cancer Institute of Emory University.
* After signing the informed consent and Health Insurance Portability and Accountability Act (HIPAA) forms, a screening evaluation will be performed. Subjects who are eligible will meet with the physical therapist and will enroll on an 8-week program of physical conditioning.
* Each patient will participate in 2-3 exercise sessions per week supervised by a physical therapist and a home exercise program. Evaluations of physical fitness will be performed before and after the 8-week exercise program. Each exercise session will be customized based on each patient's baseline fitness level. Subjects' heart rate, blood pressure, and rate of perceived exertion score will be monitored during the exercise treatment session.
* Patients' fitness at the conclusion of the physical therapy regimen will be assessed by checking for improvement in Eastern Cooperative Oncology Group (ECOG) performance status by at least 1 point from baseline and 25% improvement in the Special Forces (SF)-36 fitness scoring system.
* Decitabine will be infused according to standard of care practice with daily infusions for 5 consecutive days of a 28-day cycle for 2 cycles (1 cycle = 28 days) during the 8 week physical-conditioning period.
* Patients will be assessed by the hematology provider on a weekly basis, and adverse events/toxicities will be recorded on an ongoing basis.
* Bone marrow biopsies will be obtained at baseline, at 8 weeks, and as clinically indicated to assess for response. A sample of marrow will be collected for correlative assays coincident with the standard of care collections.
* Peripheral blood (20 mL) will be collected for correlative studies at baseline, 4 weeks and 8 weeks.

Assessment of Disease Response:

* Complete blood counts (CBC) with differential will be obtained weekly and bone marrow biopsy and aspirates will be obtained as clinically indicated to assess response to treatment.
* Active participation in the study will end 1 month after completion of the 8-week exercise/decitabine program. Thereafter, long term follow-up for survival will be performed by record review or telephone interview for patients who no longer follow-up at Winship Cancer Institute of Emory University.

Monitoring:

The study will be monitored by the Data Safety Monitoring Committee at the study institution.

Statistical Methods:

* Feasibility: Based on data showing that 50% of older fit AML patients tolerated a 4-week exercise regimen, feasibility is defined as:

  * Completion of the 8-week physical conditioning regimen/decitabine program in at least 30% of the study subjects.
  * The proportion of patients with full treatment delivery will be estimated with an exact 90% confidence interval.
* Assessment for fitness of the study population will be undertaken at 4 weeks from enrollment and conclusion of the 8-week physical therapy regimen.
* Kaplan-Meier curves will be used to estimate the distribution of time to relapse, disease-free survival, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML including de novo, secondary, or with an antecedent hematologic disorder (AHD) according to the World Health Organization (WHO) criteria
* Age ≥ 60 years
* Patient not eligible for (immediate) standard induction chemotherapy based on the opinion of the treating physician and the frailty score
* Provide signed written informed consent
* Be able to comply with study procedures and follow-up examinations
* Adequate heart function with echocardiogram demonstrating ejection fraction ≥ 45% with no evidence of systolic dysfunction
* Adequate renal and hepatic function:

  * Total bilirubin ≤ 2x institutional Upper Limit of Normal (ULN); and
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3x ULN; and
  * Serum creatinine ≤ 2 times the upper limit of normal
* ECOG performance < 4
* Patients with a history of carcinoma in remission (on no therapy or on hormonal therapy for the adjuvant treatment of breast carcinoma or prostate carcinoma) are included in the study.

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL, French-American-British [FAB] classification M3 or WHO classification of APL with t(15;17)(q22;q12)), (PML/retinoic acid receptor alpha [RARa] and variants)
* Prior treatment with decitabine for myelodysplastic syndrome (MDS) or AML
* Relapsed or refractory AML
* Rapidly doubling white cell count uncontrolled with hydroxyurea
* Coronary artery disease with angina limiting exercise capability
* Joint disease limiting exercise capability
* Investigational agent received within 30 days prior to the first dose of study drug. If received any investigational agent prior to this time point, drug-related toxicities must have recovered to Grade 2 or less prior to first dose of study drug
* Psychiatric disorders that would interfere with consent, study participation, or follow-up
* Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Any other severe concurrent disease, or serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo the proposed therapy
* No social support or inability to attend study-related visits
* Carcinoma requiring systemic chemotherapy or radiation therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Performance status | Up to 8 weeks
  ECOG performance status is assessed before, at 4 weeks and 8 weeks from start of the intervention.
Proportion of patients with 25% improvement in fitness scores | Up to 8 weeks
  Patients will be asked to answer questions on the 36-item (SF-36) fitness scoring system and the FACIT-Leu fatigue scale at baseline, 4 weeks and 8 weeks of the study.
Function | 8 weeks
  Function will be measured using the 6-meter walk test, timed Up and Go test, grip strength and lower limb strength.
Activity | 8 weeks
  Activity will be based on daily stepping activity (measured using step activity monitors), endurance (distance ambulated in 3-minutes), and duration of aerobic exercise (treadmill walking or cycling) at 50% heart rate and/or Borg score > 5.

SECONDARY OUTCOMES:
Number of patients with adverse events related to the intervention. | 8 weeks
  Toxicities will be monitored on an ongoing basis, based on review of symptoms, physical examination, and laboratory tests weekly. Adverse events (AEs) will be monitored and recorded on case report forms on an ongoing basis and will be graded using the NCI Common Toxicity Criteria (CTC) AE V. 4.
Response to treatment | 18 months
  This outcome will evaluate the response to treatment (complete response, disease-free survival [DFS], and overall survival [OS]) of the rehabilitated patients after conclusion of the 8-week program. Disease status will be assessed by a peripheral blood and bone marrow aspirate and biopsy as clinically indicated.
Quality of life and depression scores among study subjects before and after the 8-week exercise program | 8 weeks
  This outcome will evaluate changes in quality of life among study subjects before and after the 8-week exercise program, from quality of life questionnaires and depression scores.

CONTACTS AND LOCATIONS:
Overall Officials: Martha L Arellano, MD, Principal Investigator — Emory University
Locations (1):
- Winship Cancer Institute of Emory University, Atlanta, Georgia, United States